CLINICAL TRIAL: NCT07073391
Title: Laminar Circuit Motifs for Working Memory and Language Combinatorics: From Cells to Systems
Brief Title: Clinical Study of How Information Flows Across the Human Cortical Sheet Layers (Laminae), Aiming to Discover Key Principles of Laminar Circuits and Information Flow for Complex Behavior.
Acronym: LamCircuits
Status: Not yet recruiting | Type: Observational
Sponsor: Christopher I. Petkov (Other)
Collaborators: University of Minnesota (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Christopher I. Petkov, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: U01NS137991 (NIH); U01NS137991 (NIH)
Record Dates: First submitted 2025-06-30; First posted 2025-07-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neuronal Mechanisms; Laminar Circuits
Keywords: laminar array recordings; single unit recordings; cortical layers; laminar fMRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Brain tissue samples from tissue that would be clinically resected or disrupted by the patient's treatment procedure in the operating room
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Laminar Circuit Motif Observation Group: Laminar Circuit Motif Observation Cohort
  Interventions: Device: Recording with laminar arrays

INTERVENTIONS:
Device: Recording with laminar arrays — Part of the intervention is reliant on FDA approved laminar recording electrodes already available in the US. The other part will be an investigational device that is currently being considered by the FDA for an Investigational Device Exclusion.

SUMMARY:
This is a basic science study of a missing dimension of human brain function, how information flows the six layers of the brain. The research will involve neurosurgery patients and controls in laminar-resolution functional MRI at 7 Tesla during a working memory and language task. The neurosurgery patients will be involved in intracranial recordings with FDA approved electrodes capable of recording across the cortical layers, or electrodes with FDA Investigational Device Exemption. The neurosurgery patients will also be able to provide tissue samples for genomics research from tissue that would be clinically removed, resected or disrupted as part of the clinical treatment. The outcome is unprecedented insights into this missing dimension of human brain function which will help to advance biomedical science and could be crucial for developing better patient diagnostic and treatment options for a host of brain disorders where laminar information flow is disrupted but currently cannot be effectively studied.

DETAILED DESCRIPTION:
Humans are uniquely capable of combining information in novel ways to give meaning and infer unobservable causes in the environment. This ability is supported by interactions between working memory and sensory processes. When applied to language, these combinatorial processes give us the ability to reason and plan. This complex behavior is thought to be grounded in information flowing both forward and backward between cortical areas, routed through the six layered organization of the mammalian neocortex. Testing this hypothesis requires gathering information of human laminar circuits at multiple scales, from the molecular (informing the composition of local circuits) to the mesoscopic (detailing information flow within an area across laminae) and network (across areas) ones. This challenging objective has so far remained out of reach, investigating laminar circuits has been mostly confined to animal models, limiting our understanding of human complex behaviors. To break through, the investigators propose a partnership that can provide these much needed multiscale observations in 100+ neurosurgery patients and: 1) record both high-density (laminar) array recordings and subdural recordings from prefrontal and temporal cortical areas while patients conduct a task that requires the manipulation of linguistic information in working memory; 2) characterize the laminar cell-specific molecular and genetic properties of tissue sampled immediately after the recordings; and 3) scale laminar circuit insights to mesoscopic levels accessible with laminar fMRI at 7 Tesla, in the same patients undergoing electrophysiological recordings. By combining this information using a (generative) computational modeling approach, the investigators will unravel how local neural dynamics and forward and backward information passing across areas supports our ability to recombine linguistic information in working memory. The unique multiscale level information of human brain function that the investigators aim to collect will benefit efforts beyond the cognitive field, such as those oriented at understanding the biophysical processes underlying non-invasive recordings such as fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Eligible for wake DBS implantation or epilepsy/tumor/biopsy treatment procedure, within the age range of 18 and 80 years old.
* Healthy controls: can only participate in the non-invasive brain imaging study, within the age range of 18 and 80 years old.

Exclusion Criteria:

* Psychiatric disorder
* Drug addiction
* Not able to conduct an English based language task
* Not capable of being scanned with MRI (e.g., metal implants)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidate patient research participants are those requiring DBS implant, epilepsy/tumor/biopsy resection procedures that require awake treatment with craniotomy. The patients can participate in the intracranial recordings, brain imaging and tissue sampling parts of the research. Control healthy participants will only participate in the non-invasive brain imaging study with fMRI in 7 Tesla.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Observation of Laminar Circuit Motifs | From enrollment to the end of the clinical study at 5 years
  The primary objective is whether and how laminar profiles deviate from baseline under the different observational conditions: laminar fMRI, laminar array recordings and with tissue sampling genomics. A score of 0 indicates no significant deviation therefore no laminar information flow. A significant profile will indicate information flow across the cortical layers with the profile identifying which layers are involved in information flow across the cortical layers. This primary outcome will be studied individually by patients and in the cohort as a group.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Petkov, PhD, Study Director — University of Iowa

IPD SHARING:
Plan to Share IPD: No